CLINICAL TRIAL: NCT01145209
Title: A Phase II Study of Ofatumumab-Based Induction Chemoimmunotheraphy Followed by Consolidation Ofatumumab Immunotherapy in Previously Untreated Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Ofatumumab-based Induction Chemoimmunotherapy in Previously Untreated Patients With CLL/SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: University of Virginia (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100141; 10-H-0141
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Small Lymphocytic Lymphoma; CLL (Chronic Lymphocytic Leukemia)
Keywords: Arzerra; Chemoimmunotherapy; SLL; Monoclonal Antibody Therapy; CLL; Ofatumumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — fludarabine phosphate; ofatumumab; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FO Arm (fludarabine and ofatumumab) (Experimental): For patients with non-high risk FISH changes
  Interventions: Drug: Fludarabine Phosphate; Biological: Ofatumumab
- FCO Arm (fludarabine, cyclophosphamide, and ofatumumab) (Experimental): For patients with high risk FISH changes
  Interventions: Drug: Fludarabine Phosphate; Biological: Ofatumumab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given IV
  Other Names: Fludara
Biological: Ofatumumab — Given IV
  Other Names: Arzerra
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan; Neosar
  Arms: FCO Arm (fludarabine, cyclophosphamide, and ofatumumab)

SUMMARY:
Background:

- Ofatumumab was approved by the U.S. Food and Drug Administration to treat patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who have not responded to standard chemotherapy. Ofatumumab is a substance that recognizes specific types of white blood cells called B-lymphocytes, which become cancerous in CLL/SLL. Ofatumumab attaches to a molecule called CD20, which is found on the surface of B-cells, and destroys them. Previous studies have shown that ofatumumab can decrease the number of B-cells in patients with CLL/SLL who have been treated with chemotherapy, but more research is needed to determine it if can also be used to treat patients with previously untreated CLL/SLL.

Objectives:

- To determine a safe and effective dose of ofatumumab, along with chemotherapy, to treat chronic lymphocytic leukemia or small lymphocytic lymphoma.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with CLL or SLL that has not been treated with chemotherapy.

Design:

* Eligible participants will be screened with a physical exam, blood samples, lymph node and bone marrow biopsies, and imaging studies.
* Participants will be separated into 2 groups: all participants will receive ofatumumab and fludarabine, and some participants will be selected to also receive cyclophosphamide (based on results of certain blood tests).
* Participants will receive the study drugs (ofatumumab and fludarabine, and optional cyclophosphamide) by infusion for a maximum of 6 days, followed by 21 days off drug.
* Participants will have 6 cycles of treatment according to a schedule set by the study doctors, and may have their dose levels adjusted if side effects develop.
* Participants who have disease remaining after 6 cycles will receive additional ofatumumab every 2 months, starting 2 months after the end of the 6th cycle and continuing for a total of 4 doses, before entering the follow-up phase of the trial. Participants who do not have residual disease after 6 cycles will not receive additional therapy, and will immediately enter the follow-up phase of the trial.
* Participants will have a follow-up exam every 2 to 4 months for 2 years after the end of treatment, and then as required by the study doctors for as long as the study remains open. These visits will involve a full medical exam, blood samples, lymph node and bone marrow biopsies, and imaging studies.

DETAILED DESCRIPTION:
OUTLINE:

Patients with adverse interphase cytogenetics (11q22 or 17p13 deletion) receive FCO induction therapy:

* Ofatumumab is given IV on day 1 (300 mg) and day 8 (1000 mg) of course 1 and on day 1 (1000 mg) of all subsequent courses.
* Fludarabine phosphate (25mg/m2/d) and cyclophosphamide (250mg/m2/d) are given IV on days 2 through 4 of course 1 and on days 1 through 3 of all subsequent courses. Patients age 70 or older will be given reduced doses of fludarabine (20mg/m2/d) and cyclophosphamide (150mg/m2/d).
* Treatment repeats every 28 days for up to 6 courses in the absence of disease progression.

Patients without adverse interphase cytogenetics receive FO induction therapy:

* Ofatumumab is given IV on day 1 (300mg) and day 8 (1000mg) of course 1 and on day 1 (1000mg) of all subsequent courses.
* Fludarabine phosphate (25mg/m2/d) is given IV on days 2 through 6 of course 1 and on days 1 through 5 of all subsequent courses.
* Treatment repeats every 28 days for up to 6 courses in the absence of disease progression.

All patients are evaluated for minimal residual disease (MRD) by four-color flow cytometric analysis of the peripheral blood after completion of FO or FCO induction therapy, and are subsequently stratified into two groups:

* Patients who are MRD-positive and without evidence of disease progression proceed to consolidation therapy beginning approximately 5 months after completion of induction therapy, consisting of ofatumumab (1000mg) given IV on day 1 of all courses. Treatment repeats every 2 months for up to 4 courses in the absence of disease progression. Patients are followed clinically 2 and 6 months after the last dose of ofatumumab is given, and then every 6 months thereafter.
* Patients who are MRD-negative and without evidence of disease progression are followed clinically every 4 months for 1 year and every 6 months thereafter.

ELIGIBILITY:
* INCLUSION CRITERIA:

Histologically confirmed CLL or SLL as defined by the following:

* B-lymphocytosis greater than 5000 cells/micro L (may be less than 5000 cells/micro L if lymphadenopathy is present with histologic confirmation of lymph node involvement by SLL).
* Immunophenotypic profile consistent with CLL as demonstrated by flow cytometry
* Appropriate immunophonotype (CD5/19/23+)
* Clonality of lymphocytosis confirmed by flow cytometry
* large lymphocytes less than 55 % of blood lymphocytes

Active disease as defined by at least one of the following:

* Weight loss greater than or equal to10 percent within the previous 6 months
* Extreme fatigue
* Fevers of greater than 100.5 degree F for greater than or equal to 2 weeks without evidence of infection
* Night sweats for more than one month without evidence of infection
* Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
* Massive or progressive splenomegaly
* Massive nodes or clusters or progressive lymphadenopathy
* Progressive lymphocytosis with an increase of greater than 50% over a 2 month period, or an anticipated doubling time of less than 6 months 0

Measurable disease (defined as two dimensional disease on imaging or quantifiable leukemic disease).

Ages 18 and over.

EXCLUSION CRITERIA:

Prior monoclonal antibody therapy with agents having anti-CLL activity

Prior cytotoxic chemotherapy with agents having anti-CLL activity (Fludarabine, Cyclophosphamide, Bendamustine, Chlorambucil)

Transformed CLL

Active autoimmune hemolytic anemia or thrombocytopenia

Any medical condition that requires the chronic use of corticosteroids

Active or latent Hepatitis B infection

HIV infection

Severe chronic obstructive pulmonary disease, severe cardiac disease, or other uncontrolled medical condition that would, in the opinion of the principal investigator, place the subject at an unreasonable risk of life-threatening adverse events due to chemoimmunotherapy

ECOG performance status 3 or worse

Creatinine greater than or equal to 2 mg/dL or creatinine clearance less than or equal to 30 mL/min

Bilirubin greater than or equal to 2 mg/dL or active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment)

Female patients: Current pregnancy or unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential or currently breastfeeding. Male patients who are unwilling to follow the contraception requirements described in this protocol.

Psychiatric illness/social situations that would limit the patient s ability to tolerate and/or comply with study requirements.

Unable to understand the investigational nature of the study or give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07-01; Primary Completion 2017-10-31 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inhye Ahn, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahn I, Farooqui M, Lee YS, Marti G, Soto S, Tian X, Stetler-Stevenson M, Yuan CM, Maric I, Wiestner A. Risk-Adapted Induction and Maintenance with Ofatumumab in Previously Untreated Patients with Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL). Blood 2015 126(23):1750-1750.
- [Background] Desai S, Mo C, Gaglione EM, Yuan CM, Stetler-Stevenson M, Tian X, Maric I, Wake L, Farooqui MZ, Drinkwater DC, Soto S, Valdez J, Hughes TE, Nierman P, Lotter J, Marti GE, Pleyer C, Sun C, Superata J, Nichols C, Herman SEM, Lindorfer MA, Taylor RP, Wiestner A, Ahn IE. Risk-adapted, ofatumumab-based chemoimmunotherapy and consolidation in treatment-naive chronic lymphocytic leukemia: a phase 2 study. Leuk Lymphoma. 2021 Aug;62(8):1816-1827. doi: 10.1080/10428194.2021.1888379. Epub 2021 Mar 2. PMID 33653216
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-H-0141.html

RESULTS

PARTICIPANT FLOW:
Groups:
- FCO Arm (Fludarabine, Cyclophosphamide, and Ofatumumab): Fludarabine, cyclophosphamide, and ofatumumab for patients with high-risk FISH changes
- FO Arm (Fludarabine and Ofatumumab): Fludarabine and ofatumumab for patients with non-high-risk FISH changes
Period: Overall Study
Arm/Group | FCO Arm (Fludarabine, Cyclophosphamide, and Ofatumumab) | FO Arm (Fludarabine and Ofatumumab)
Started | 13 | 19
Completed | 10 | 18
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) requiring first-line therapy for CLL or SLL
Groups:
- Total: Total of all reporting groups
Arm/Group | FO Arm (Fludarabine and Ofatumumab) | FCO Arm (Fludarabine, Cyclophosphamide, and Ofatumumab) | Total
Number analyzed (Participants) | 19 | 13 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 8 | 23
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 17 | 10 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate 2 Years After Initiation of Induction Therapy
Description: Death or disease progression defined by the 2008 IWCLL guideline as follows;
  * Greater than or equal to 50% increase in the SPD of at least 2 lymph nodes (at least one node must be greater than or equal to 2 cm); appearance of any new lymph nodes on physical examination or imaging
  * Greater than or equal to 50% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margin or CT scan or appearance of palpable hepatomegaly or splenomegaly, which was not previously present
  * Greater than or equal to 50% increase in the absolute number of circulating lymphocytes to at least 5000/ul
  * Transformation to a more aggressive histology
  * Occurrence of any cytopenia attributable to CLL. After treatment: the progression of any cytopenia (unrelated to autoimmune cytopenia), as documented by a decrease of Hb levels by more than 20 g/L (2 g/dL) or to less than 100 g/L (10 g/dL), or by a decrease of platelet counts by more than 50% or to les
Time Frame: 2 years
Population: The analyses included only those subjects who completed the induction period.
Measure: Count of Participants; unit: Participants
Groups:
- FO Arm: Fludarabine and ofatumumab for patients with non-high-risk FISH changes
- FCO Arm: Fludarabine, cyclophosphamide, and ofatumumab for patients with high-risk FISH changes
Arm/Group | FO Arm | FCO Arm
Number analyzed (Participants) | 18 | 10
Participants | 14 | 9

2. Secondary Outcome: Number of Grade 3 and 4 Treatment Related Adverse Events
Description: Number of Grade 3 and 4 treatment related adverse events as defined by CTCAE version 3.0 criteria.
  CTCAE (Common Terminology Criteria for Adverse Events) provides a list of adverse event (AE) terms commonly reported. Each AE term is defined and accompanied by a grading scale that indicates the severity of the AE. The CTCAE v3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 is a Mild AE; Grade 2 is a Moderate AE; Grade 3 is a Severe AE; Grade 4 is a Life-threatening or disabling AE; and Grade 5 is a Death related to AE
Time Frame: 2 years
Population: All patients included in safety analysis. It was pre-specified to recombine Arms/Groups for this assessment and report irrespective of randomized group.
Measure: Number; unit: Number of Grade 3 and Grade 4 AEs
Groups:
- FO + FCO Arms: Participants received Fludarabine and ofatumumab for patients with non-high-risk FISH changes or Fludarabine, cyclophosphamide, and ofatumumab for patients with high-risk FISH changes.
Arm/Group | FO + FCO Arms
Number analyzed (Participants) | 32
Number of Grade 3 and Grade 4 AEs
  Neutropenia Grade 3 | 4
  Thrombocytopenia Grade 3 | 2
  Nausea Grade 3 | 1
  Infusion reaction Grade 3 | 1
  Neutropenia Grade 4 | 17
  Lymphopenia Grade 4 | 2

3. Secondary Outcome: Participants With Minimal Residual Disease (MRD) Negativity
Description: Participants with minimal residual disease (MRD) negativity following the completion of induction chemoimmunotherapy.
Time Frame: 2 years
Population: The analyses included only those subjects who completed the induction period.
Measure: Count of Participants; unit: Participants
Arm/Group | FO ARM | FCO ARM
Number analyzed (Participants) | 18 | 10
Participants | 4 | 6

4. Secondary Outcome: Participants With MRD Negativity at the Completion of Consolidation Immunotherapy Who Failed to Achieve MRD Negativity
Description: Participants with MRD negativity at the completion of consolidation immunotherapy who failed to achieve MRD negativity following completion of induction chemoimmunotherapy
Time Frame: 2 years
Population: Participants who achieved MRD negativity at the completion of consolidation immunotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | FO Arm | FCO Arm
Number analyzed (Participants) | 14 | 4
Participants | 14 | 4

5. Secondary Outcome: Participants With Complete Response Rates Following Induction Chemoimmunotherapy.
Description: Participants with complete response rates to induction chemoimmunotherapy.
  Criteria for complete response (CR): CR requires all of the following:
  * Peripheral blood lymphocytes < 4000/uL
  * Absence of significant lymphadenopathy by physical examination and appropriate radiographic techniques (CT or MRI). All lymph nodes must have regressed to <=1.5cm in greatest diameter
  * Absence of hepatomegaly or splenomegaly by physical examination, or appropriate radiographic techniques. Spleen, if enlarged before therapy must have regressed in size and must not be palpable by physical exam.
  * Absence of constitutional symptoms
  * Normal CBC, defined as: - Polymorphonuclear cells ≥ 1,500/uL - Platelets > 100,000/uL (untransfused) - Hemoglobin > 11 g/dL (untransfused)
  * Bone marrow biopsy demonstrates normal cellularity for age, with less than 30% of nucleated cells being lymphocytes. Lymphoid nodules should be absent
Time Frame: 2 years
Population: The analyses included only those subjects who completed the induction period.
Measure: Count of Participants; unit: Participants
Groups:
- FCO Arms: Fludarabine, cyclophosphamide, and ofatumumab for patients with high-risk FISH changes
Arm/Group | FCO Arms | FO Arm
Number analyzed (Participants) | 10 | 18
Participants | 6 | 2

6. Secondary Outcome: Participants Overall Response Rates Following Induction Chemoimmunotherapy.
Description: Participants with complete response rates to induction chemoimmunotherapy.
  Criteria for complete response (CR) requires all of the following: Peripheral blood lymphocytes < 4000/uL. No significant lymphadenopathy. Lymph nodes regressed to <=1.5cm. No hepatomegaly or splenomegaly. Spleen, if enlarged before therapy must have regressed in size and not be palpable. Absence of constitutional symptoms. Bone marrow biopsy demonstrates normal cellularity for age, with less than 30% of nucleated cells being lymphocytes. No lymphoid nodules.
  Criteria for partial response (PR) requires at least one element of an abnormal CBC and at least one of the following: ≥ 50% decrease in peripheral blood lymphocyte count; ≥ 50% reduction in the sum of the products of lymph nodes up to 6 nodes or nodal masses. No new sites or increase in size of nodes; ≥ 50% reduction in pathologic enlargement of the liver and/or spleen by 50%.
Time Frame: 2 years
Population: The analyses included only those subjects who completed the induction period.
Measure: Count of Participants; unit: Participants
Groups:
- FCO Arm: Participants received Fludarabine, cyclophosphamide, and ofatumumab for patients with high-risk FISH changes.
Arm/Group | FCO Arm | FO Arm
Number analyzed (Participants) | 10 | 18
Participants
  Complete Response | 6 | 2
  Partial Response | 4 | 16

7. Secondary Outcome: Participants Overall Survival Rate After Initiation of Induction Chemoimmunotherapy
Description: Participants overall survival rate 2 years after initiation of induction chemoimmunotherapy
Time Frame: Up to 2 years
Population: The analyses included only those subjects who completed the induction period.
Measure: Count of Participants; unit: Participants
Arm/Group | FO Arm | FCO Arm
Number analyzed (Participants) | 18 | 10
Participants
  Alive | 18 | 10
  Deaths | 0 | 0

8. Secondary Outcome: Median Relationship of CD20 Expression With MRD Negativity Rate
Description: Median relationship of biomarker, CD20 expression with MRD negativity clinical response rate. Flow cytometry was use to quantified surface CD20 on peripheral blood.
Time Frame: 2 years
Population: The analyses included only those subjects who completed the induction period. It was pre-specified to have arms/groups recombine for this assessment and report irrespective of randomized group.
Measure: Median (Full Range); unit: sites per cell
Groups:
- Minimal Residual Disease (MRD) Positivity: Participants with Minimal Residual Disease (MRD) positivity following induction therapy received consolidation Ofatumumab for 4 cycles.
- Minimal Residual Disease (MRD) Negativity: No additional therapy received for participants that had Minimal Residual Disease (MRD) negativity.
Arm/Group | Minimal Residual Disease (MRD) Positivity | Minimal Residual Disease (MRD) Negativity
Number analyzed (Participants) | 18 | 9
sites per cell | 10247 [2336 to 20956] | 15131 [3323 to 55488]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Based on CTCAE version 4 for non-hematologic toxicities and 2008 IWCLL guidelines for hematologic toxicities
Groups:
- FCO (Fludarabine, Cyclophosphamide, and Ofatumumab): Fludarabine, cyclophosphamide, and ofatumumab for patients with high-risk FISH changes
- FO (Fludarabine and Ofatumumab): Fludarabine and ofatumumab for patients with non-high-risk FISH changes
Arm/Group | FCO (Fludarabine, Cyclophosphamide, and Ofatumumab) | FO (Fludarabine and Ofatumumab)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/19
Serious Adverse Events (participants affected / at risk) | 4/13 | 4/19
Other Adverse Events (participants affected / at risk) | 13/13 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FCO (Fludarabine, Cyclophosphamide, and Ofatumumab) (N=13) | FO (Fludarabine and Ofatumumab) (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FCO (Fludarabine, Cyclophosphamide, and Ofatumumab) (N=13) | FO (Fludarabine and Ofatumumab) (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Chest pain (Cardiac disorders) | 2 | 0
Dizziness (Cardiac disorders) | 4 | 4
Dyspnea (Cardiac disorders) | 3 | 1
Oedema peripheral (Cardiac disorders) | 1 | 2
Ear hemorrhage (Ear and labyrinth disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 6
Oral candidiasis (Gastrointestinal disorders) | 0 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Chills (General disorders) | 2 | 3
Decreased appetite (General disorders) | 0 | 1
Fatigue (General disorders) | 8 | 11
Flushing (General disorders) | 1 | 2
Hyperhidrosis (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 2
Night sweats (General disorders) | 1 | 1
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Hepatitis viral (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 5 | 6
Rhinitis allergic (Immune system disorders) | 2 | 2
Lung infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 9
Urinary tract infection (Infections and infestations) | 0 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Phlebitis (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Hemoglobin (Investigations) | 2 | 0
Haptoglobin (Investigations) | 0 | 1
International normalized ratio increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 9 | 13
Platelet count decreased (Investigations) | 2 | 2
White blood cell count increased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Osteopenia (Metabolism and nutrition disorders) | 1 | 0
Pica (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abnormal dreams (Nervous system disorders) | 2 | 0
Cerebral ischemia (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Confusional state (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 6
Insomnia (Nervous system disorders) | 1 | 7
Neuralgia (Nervous system disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT01145209/Prot_SAP_000.pdf